CLINICAL TRIAL: NCT01999894
Title: An Open-label Extension Study of the Safety and Tolerability of Memantine in Pediatric Patients With Autism
Brief Title: Open-label Study of Safety and Tolerability of Memantine in Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEM-MD-67
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-01

CONDITIONS: Autism; Pediatric Autism
Keywords: Namenda; Autism; Memantine; Pediatric; Forest Laboratories
MeSH Terms: conditions — Autistic Disorder | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Experimental): Once daily oral administration of memantine for 48 weeks: 6-week double-blind dose-titration period followed by a 42-week maintenance period.
  Interventions: Drug: Memantine HCl

INTERVENTIONS:
Drug: Memantine HCl — Memantine extended release 3- and 6-mg capsules; dose ranging 3 - 18 mg/day; weight based dosing in 4 weight groups; oral administration. Dosing is once daily for 48 weeks.
  Other Names: Namenda; Namenda XR

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of memantine in the treatment of autism in pediatric patients.

DETAILED DESCRIPTION:
This is a 48-week multicenter extension study comprised of a 6-week double-blind dose-titration period followed by a 42-week open-label maintenance period.

In the Forest autism trials conducted in children ages 6-12, dosing with an extended release formulation of memantine was weight-based. These weight based dose limits were selected to ensure exposure in terms of area under the curve (AUC) was less than the predefined limit of 2100 ng∙h/mL that represented a 10-fold lower exposure than observed at the NOAEL (No observed adverse effect level) of 15 mg/kg/day in juvenile rats.

The weight-based dose limits in these studies were as follows:

* Group A: ≥ 60 kg; max 15 mg/day
* Group B: 40-59 kg; max 9 mg/day
* Group C: 20-39 kg; max 6 mg/day
* Group D: < 20 kg; max 3 mg/day

ELIGIBILITY:
Inclusion Criteria:

* Completed lead-in study MEM-MD-57A (NCT00872898)
* A knowledgeable caregiver capable of providing reliable information about the patient's condition, able to attend all clinic visits with the patient

Exclusion Criteria:

* Patients with a concurrent medical condition that might interfere with the conduct of the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2009-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim Katz, PhD, Study Director — Forest Laboratories
Locations (19):
- United States (19):
  - Forest Investigative Site 005, Phoenix, Arizona
  - Forest Investigative Site 003, Sacramento, California
  - Forest Investigative Site 021, San Francisco, California
  - Forest Investigative Site 026, Santa Ana, California
  - Forest Investigative Site 020, Santa Ana, California
  - Forest Investigative Site 002, Stanford, California
  - Forest Investigative Site 024, Jacksonville Beach, Florida
  - Forest Investigative Site 007, St. Petersburg, Florida
  - Forest Investigative Site 014, Hoffman Estates, Illinois
  - Forest Investigative Site 023, Naperville, Illinois
  - Forest Investigative Site 010, Indianapolis, Indiana
  - Forest Investigative Site 025, Cambridge, Massachusetts
  - Forest Investigative Site 011, Toms River, New Jersey
  - Forest Investigative Site 006, Voorhees Township, New Jersey
  - Forest Investigative Site 017, Manhasset, New York
  - Forest Investigative Site 013, Cleveland, Ohio
  - Forest Investigative Site 015, Cleveland, Ohio
  - Forest Investigative Site 001, Columbus, Ohio
  - Forest Investigative Site 019, Oklahoma City, Oklahoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who completed the lead-in study MEM-MD-57A (NCT00872898) were eligible to enroll in this study. A total of 19 study centers in the United States enrolled patients.
Pre-assignment Details: Patients receiving placebo in the lead-in study underwent a double-blind up-titration targeting same weight-based dose assigned at lead-in study. Patients receiving a stable dose of active were not re-titrated but double-blind was maintained. Patients who were not dosed for more than 3 days between the studies underwent an open-label titration.
Groups:
- Memantine: Once daily oral administration of memantine extended release. Memantine - 3mg and 6mg capsules, dose ranging 3 - 18 mg/day; weight based dosing in 4 weight groups.
Period: Overall Study
Arm/Group | Memantine
Started | 102
Completed | 66
Not Completed | 36
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 5
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 10
Not completed — Other Reason | 3
Not completed — Inclusion/exclusion criteria not met | 1

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years]
  Years | 9.1 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 87
Race/Ethnicity, Customized [Number; unit: participants]
  White | 86
  Black | 2
  Asian | 9
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 1
  Other | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 11
  Non-Hispanic or Latino | 91
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: Number of patients who experienced one or more TEAEs during the study
Time Frame: From Visit 1 (Week 1) to 30 days after Visit 8 (Week 48)
Population: The Safety Population consists of 102 enrolled patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Memantine
Number analyzed (Participants) | 102
participants | 85

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 40 month period from November 2009 to March 2013 at 19 study sites in the US.
Groups:
- Placebo to Memantine: Patients who received placebo during the double-blind lead-in study, were titrated to Memantine during a 6-week lead-in to 42 weeks of Open Label Memantine - Once daily oral administration of memantine extended release. Memantine - 3mg and 6mg capsules, dose ranging 3 - 18 mg/day; weight based dosing in 4 weight groups.
- Memantine to Memantine: Patients who received Memantine during the double-blind lead-in study continued to receive Memantine during a 6-week lead-in, followed by 42 weeks of Open Label Memantine - Once daily oral administration of memantine extended release. Memantine - 3mg and 6mg capsules, dose ranging 3 - 18 mg/day; weight based dosing in 4 weight groups.
Arm/Group | Placebo to Memantine | Memantine to Memantine
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/52
Other Adverse Events (participants affected / at risk) | 37/50 | 37/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Memantine (N=50) | Memantine to Memantine (N=52)
Lobar pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to Memantine (N=50) | Memantine to Memantine (N=52)
Constipation (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 6 | 2
Irritability (General disorders) | 2 | 5
Pyrexia (General disorders) | 1 | 5
Seasonal allergy (Immune system disorders) | 7 | 2
Nasopharyngitis (Infections and infestations) | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 10
Weight increased (Investigations) | 5 | 4
Headache (Nervous system disorders) | 4 | 3
Psychomotor hyperactivity (Nervous system disorders) | 3 | 3
Aggression (Psychiatric disorders) | 5 | 3
Agitation (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Ear Infection (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 3 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 4
Bronchitis (Infections and infestations) | 3 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Stereotypy (Psychiatric disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.